CLINICAL TRIAL: NCT07302737
Title: Accuracy of Different Biomarkers for Predicting Delirium in Older Adults With Heart Failure
Brief Title: Delirium and Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD195/2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Delirium Confusional State
Keywords: Heart failure; delirium; older adults
MeSH Terms: conditions — Heart Failure; Confusion; Delirium | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: hospitalized older patients with heart failure and delirium
  Interventions: Other: Comprehensive Geriatric Assessment; Other: the Confusion Assessment Method (CAM test) or CAM-ICU; Other: Delirium Rating Scale - Revised-98; Diagnostic Test: blood biomarkers
- controls: age and gender matched heart failure older patients without delirium
  Interventions: Other: Comprehensive Geriatric Assessment; Other: the Confusion Assessment Method (CAM test) or CAM-ICU; Diagnostic Test: blood biomarkers

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — multidimensional assessment of cognition, physical, function, mood, social status of the participants
Other: the Confusion Assessment Method (CAM test) or CAM-ICU — standardized tool designed to quickly and accurately diagnose delirium by assessing four key features: acute mental change, inattention, and either disorganized thinking or altered consciousness. The original CAM is used for communicative patients on general wards, relying on conversation, while the CAM-ICU is adapted for critically ill, often non-verbal patients in the ICU, using non-verbal tasks and sedation scales. By providing a rapid, reliable method for identifying this often-missed condition, both tools trigger crucial medical interventions, helping to mitigate delirium's serious risks, including longer hospital stays, long-term cognitive decline, and increased mortality.
Other: Delirium Rating Scale - Revised-98 — The Delirium Rating Scale-Revised-98 (DRS-R-98) is a standardized, expert-rated clinical tool designed specifically to measure the severity of delirium and help distinguish it from other psychiatric disorders, such as dementia, depression, and schizophrenia. Unlike the CAM/CAM-ICU, which provides a simple "yes/no" diagnosis, the DRS-R-98 quantifies how severe a patient's delirium is at a given point in time and tracks changes in that severity over the course of the illness
  Groups: cases
Diagnostic Test: blood biomarkers — complete blood count(to obtain systemic inflammatory index) ,triglyceride (TG) and glucose, Liver and kidney function tests and serum electrolytes level

SUMMARY:
Biomarkers such as Systemic Immune-Inflammation Index (SII) and TG/Glucose Ratio (TyG) have shown promise in predicting delirium, reflecting the roles of inflammation and metabolic disturbances in its pathophysiology. This study aims to compare the predictive value of SII and the TyG ratio among other chemical and physiological biomarkers for diagnosing delirium and detecting its severity in older adults with heart failure. These biomarkers reflect different pathophysiological pathways implicated in delirium, including inflammation, cardiovascular stress, and metabolic dysfunction. By evaluating their individual and combined predictive abilities, this research seeks to identify potential tools for early identification of patients at high risk for delirium

ELIGIBILITY:
Inclusion Criteria:

Heart failure stage C

Exclusion Criteria:

1. cognitive impairment
2. Major Neurological Conditions: (e.g., stroke, traumatic brain injury).
3. Hematological diseases that affect platelet, neutrophil, and lymphocyte counts.
4. Cardiogenic Shock
5. Sepsis
6. Ongoing Treatment with Immunosuppressants, or corticosteroids

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospitalized older adults with heart failure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
the sensitivity and specificity of different biomarkers of delirium in heart failure older patient | Within 24 hours of hospital admission
  assess sensitivity and specificity of the systemic inflammatory index (SII), Rate Pressure Product (RPP), and TG/glucose ratio in predicting delirium

SECONDARY OUTCOMES:
in hospital morbidity | From enrollment to the hospital discharge about 6 weeks
  follow up cohort for possible complications like acute kidney injury, infections, or adverse drug events
In hospital mortality | From enrollment to hospital discharge about 6 weeks
  cohort follow up throughout hospital course and mortality recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided